CLINICAL TRIAL: NCT06998238
Title: The Interplay Between Androgens, Insulin, and Adipose Tissue Metabolism
Brief Title: Evaluating the Influence of Diet-induced Weight Loss on Fat (Adipose) Tissue's Insulin Sensitivity and Testosterone Synthesis in Women With Overweight or Obesity, Insulin Resistance, and Hyperandrogenemia
Acronym: WAIST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Elizabeth Jane Parks, Professor, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2095704
Record Dates: First submitted 2025-02-24; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-03

CONDITIONS: Overweight and Obesity; Hyperandrogenemia; Insulin Resistance
Keywords: Insulin resistance; Hyperandrogenemia; Weight loss; Mediterranean Diet; Women; Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dietary intervention (Experimental): Group receiving the study diet and nutrition counseling.
  Interventions: Behavioral: Mediterranean-based, carbohydrate restricted, calorie reduced diet
- Control (No Intervention): Group that performs repeat measures over the span of 8 weeks without any intervention or influence from study team in the interim.

INTERVENTIONS:
Behavioral: Mediterranean-based, carbohydrate restricted, calorie reduced diet — Dietary intervention - calorie reduced (300-500 kcal/day below estimated energy needs), carbohydrate restricted (<100 grams of available carbohydrates per day), Mediterranean-based (high fat diet with an emphasis on the addition of healthy fats - nuts, avocados, olive oil, increasing whole grains, increasing fruit and vegetables, replacing red meats with fish and poultry, reducing dairy, and reducing added sugars) diet.
  Arms: Dietary intervention

SUMMARY:
The investigators will measure plasma concentrations of the hormones insulin and testosterone as well as measures of insulin sensitivity in women with overweight or obesity who have insulin resistance (IR). Women who meet these criteria that also have elevated total or free testosterone will be eligible to participate in the diet intervention. The dietary intervention is designed to produce a 5% reduction in starting body weight to test whether weight loss will acutely lower fasting insulin and testosterone concentrations.

DETAILED DESCRIPTION:
The investigators will measure the efficacy of a diet-induced weight loss intervention to reduce blood concentrations of the hormone's insulin and testosterone over the course of 2 months in women who have overweight or obesity and evidence of IR. Women meeting the eligibility criteria that have biochemical evidence or clinical manifestations of hyperandrogenemia (HA), or elevated blood androgens - testosterone or free testosterone - will be eligible for the dietary intervention arm of the study. A Mediterranean-based, calorie reduced, carbohydrate restricted diet will be employed to produce a 5% weight loss over the 8 weeks of the intervention. Participants will be provided with a full menu of meals and snacks for 4 of the 8 weeks in the study and will meet with a registered, licensed dietitian routinely for nutrition counseling and to ensure dietary compliance. Those in the dietary intervention will undergo 6 clinical visits at the Clinical and Translational Science's Unit whereas the control group (no dietary intervention or nutrition counseling) will undergo 2 clinical visits. Of the 6 study visits, 4 will include an adipose tissue biopsy and an oral glucose tolerance test. All visits will include DEXA measurement of body composition and collection of fasting blood samples. The control group's 2 study visits will occur at the start and end of the 8-week period and will include all study measurements (i.e., adipose tissue biopsies, oral glucose tolerance tests, DEXA scans, and fasting blood samples). Adipose tissue samples will be cultured and used to assess adipose-level insulin sensitivity. Area under the curve for insulin, glucose, and non-esterified fatty acids (NEFA) will be calculated from the samples collected during the oral glucose tolerance test. Additionally, the fasting HOMA-IR, Matsuda Index, QUICKI value, 2-hour blood glucose concentration, and NEFA suppression will be measured during the oral glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Women (female sex, premenopausal)
* Age 21-45y
* Overweight/obesity with BMI ≥25.0 or ≤50.0 kg/m2
* Prediabetic (fasting glucose between 100-125 mg/dL,HbA1c between 5.7-6.4%, blood glucose ≥ 140 mg/dL, but ≤ 200 mg/dL at 2 hours into OGTT) or diabetic with a fasting glucose <200 mg/dL, stably treated with metformin for 2 months or longer
* Alternatively: if not prediabetic as evidenced by abnormal fasting blood glucose or glucose tolerance, evidence of insulin resistance such as fasting insulin value ≥ 10 µU/mL, elevated HOMA-IR or elevated QUICKI may be substituted

  o Prediabetes and diabetes are associated with insulin resistance and excess body weight. Our study seeks to improve impaired insulin signaling through weight loss from dietary restriction. Therefore, insulin resistance in the presence of normal glucose tolerance may still be improved through this intervention.
* Plasma testosterone concentration <200 ng/dL, as measured at screening visit
* Weight stable: No fluctuations in body weight of greater than 4 kg in the last 2 months (see exclusion criteria for undergoing weight loss)
* Presence of central (android) obesity as defined by WHR > 0.8 or waist circumference > 80 cm
* No use or active use of hormonal contraceptives (IUD, oral contraceptive pill, Nexplanon)

  o Hormonal contraceptives are not expected to alter the outcomes of this study; therefore, their use is not prohibited. However, it is not a requirement that women use hormonal contraception to be part of this study.
* Willingness to consume a defined diet (Intervention arm - Weight loss)

Exclusion Criteria:

* Pregnant or trying to become pregnant
* Postmenopausal as testosterone naturally increases with menopause
* BMI of <25.0 or >50.0 kg/m2
* Use of tobacco, cannabis, or other recreational drug products.

  o Tobacco and other recreational drugs products are excluded as they known to increase adipose lipolysis. Cannabis products are excluded as they are fat soluble compounds and could alter the adipose gene and protein expression.
* Taking medications known to affect adipose tissue metabolism (steroids, niacin)
* Use of antiandrogen medications (spironolactone, flutamide, finasteride) within the last 3 months o These medications are designed to lower testosterone concentrations.
* Already undergoing weight loss. o As this study is investigating the impact of weight loss, the goal is to obtain samples before and after weight loss (intervention arm) or during weight stability (control arm).
* Diagnosis of congenital adrenal hyperplasia, or Cushing syndrome o These conditions are associated with significantly high androgens in need of medical treatment.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-01-07 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in fasting hormone concentrations. | Day 0, day 7, day 14, day 28, day 42, and day 56 for the intervention group and day 0 and day 56 for the control group.
  Fasting insulin (µU/mL) will be measured and compared to baseline values. Samples are sent to an external CLIA-compliant lab (Quest Diagnostics) for analysis.
Change in fasting hormone concentrations. | Day 0, day 7, day 14, day 28, day 42, and day 56 for the intervention group and day 0 and day 56 for the control group.
  Fasting testosterone (ng/dL) will be measured and compared to baseline values. Samples are sent to an external CLIA-compliant lab (Quest Diagnostics) for analysis.
Change in body weight (kg). | Day 0, day 7, day 14, day 28, day 42, and day 56 for the intervention group and day 0 and day 56 for the control group.
  Change from baseline values will be measured using a calibrated, standard, clinical scale.
Change in fasting blood biochemistries. | Day 0, day 7, day 14, day 28, day 42, and day 56 for the intervention group and day 0 and day 56 for the control group.
  Fasting SHBG (nmol/L) will be measured and compared to baseline values. Samples are sent to an external CLIA-compliant lab (Quest Diagnostics) for analysis.

SECONDARY OUTCOMES:
Change in whole body insulin sensitivity. | Day 0, day 14, day 28, day 56 for the intervention group and day 0 and day 56 for the control group.
  Participants will undergo an oral 75-gram glucose tolerance test. Insulin sensitivity will be assessed using HOMA-IR. This insulin sensitivity index is calculated as [(fasting insulin (µU/mL) x fasting glucose (mg/dL))/405].
Indirect measure of change in adipose insulin sensitivity. | Day 0, day 14, day 28, day 56 for the intervention group and day 0 and day 56 for the control group.
  Change will be calculated relative to the fasting value as the percent suppression of free fatty acids in response to the oral glucose tolerance test. Plasma free fatty acids are measured in mmol/L.
Direct measure of change in adipose insulin sensitivity. | Day 0, day 14, day 28, day 56 for the intervention group and day 0 and day 56 for the control group.
  Abdominal subcutaneous adipose tissue (~1 gram) is collected via biopsy. Primary cells are cultured. After differentiation to fully mature adipocytes, the cells are cultured in 1 of 6 media conditions - standard (10 nM insulin, 0 ng/dL testosterone), hyperinsulinemic (100 nM insulin, 0 ng/dL testosterone), hyperinsulinemic and low testosterone (20 ng/dL), hyperinsulinemic and high testosterone (40 ng/dL), standard and low testosterone, standard and high testosterone. Following 10 days of media treatment, adipocyte insulin sensitivity is assessed via a lipolysis assay. This assay measures the release of free fatty acid (mmol/L) from adipocytes in response to cAMP and the subsequent suppression when treated with insulin.
Change in measures of biochemical hyperandrogenemia. | Day 0, day 7, day 14, day 28, day 42, and day 56 for the intervention group and day 0 and day 56 for the control group.
  Fasting free testosterone concentrations (as a percentage (%) of total testosterone) will be estimated. Values will be compared to baseline.
Change in body composition. | Day 0, day 7, day 14, day 28, day 42, and day 56 for the intervention group and day 0 and day 56 for the control group.
  Absolute (kg) and relative (percent of total body mass) fat-free and fat mass are measured using a DEXA at each study visit and compared to baseline values.
Change in average blood glucose concentrations. | Day 0 and day 56 for both the intervention and the control groups.
  Change in HbA1c % will be measured and compared to baseline values. Samples are sent to an external, CLIA compliant lab (Quest Diagnostics) for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Parks, PhD, Principal Investigator — University of Missouri-Columbia; Jean Ricci Goodman, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon reasonable request to study's primary investigator, Elizabeth J. Parks, PhD.